CLINICAL TRIAL: NCT05945186
Title: Design Validation Hemodynamic Study of New Kendall SCD SmartFlow Compression System With Cardinal Health Element Compression Sleeves
Brief Title: Design Validation Hemodynamic Study of New Kendall SCD SmartFlow Compression System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cardinal Health (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 450.30
Record Dates: First submitted 2023-07-06; First posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Hemodynamics
Keywords: Hemodynamics; Blood Flow

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single Arm (Experimental): Baseline blood flow (hemodynamic) measurements will be obtained via ultrasound for all enrolled subjects. Following baseline measurements, compression will be applied and blood flow (hemodynamic) measurements will be repeated via ultrasound.
  Interventions: Device: Intermittent Pneumatic Compression (IPC)(Kendall SCD SmartFlow™ compression system with Cardinal Health Element compression sleeves)

INTERVENTIONS:
Device: Intermittent Pneumatic Compression (IPC)(Kendall SCD SmartFlow™ compression system with Cardinal Health Element compression sleeves) — External intermittent pneumatic compression (IPC) systems are applied to subject legs and comprise of a controller, associated tubing set and single patient use disposable leg sleeves. The disposable sleeves are latex free and contain air bladder(s) that are inflated by the controller to provide compression to the legs/feet. These devices are designed to increase venous blood flow in at risk patients in order to help prevent Venous ThromboEmbolism (VTE), including Deep Vein Thrombosis (DVT) and Pulmonary Embolism (PE).

SUMMARY:
This study is being conducted to evaluate the hemodynamic performance (i.e. flow of blood) in the legs using the new Kendall SCD SmartFlow™ compression system with Cardinal Health Element compression sleeves.

DETAILED DESCRIPTION:
This study is being conducted to evaluate hemodynamic performance using the new Kendall SCD SmartFlow™ compression system with Cardinal Health Element compression sleeves. The study is intended to confirm the system's ability to increase venous blood flow over baseline as measured by blood velocity, time average mean velocity and total volume flow, in both the femoral and popliteal veins.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be ≥18 years and ≤ 89 years of age.
* Subject must be able to speak and read English.
* Subject must have both legs fully intact (cannot be an amputee) with normal function.
* Subject must be able to commit to the full study duration (approximately 1-2 hours of uninterrupted time).
* Subject legs must fit into the provided knee length compression sleeves (<32").
* Subject must give written informed consent.

Exclusion Criteria:

* Subject is currently pregnant or breastfeeding.
* Subject has a positive COVID history within the previous 6 months.
* Subject presents with

  * - local leg condition with which the sleeves would interfere such as dermatitis, vein ligation (immediate post-operative), gangrene, recent skin graft, or any other open wound
  * - arteriosclerosis or other ischemic vascular diseases as indicated by absence of pedal pulses and/or history of intermittent claudication with positive pain response
  * - edema of legs or pulmonary edema from congestive heart failure
  * - deformity of the leg
  * - current Deep Vein Thrombosis as identified during baseline clinical screening
  * - recent or old Deep Vein Thrombosis as identified during baseline clinical screening
  * - reflux in the superficial or deep veins
  * - history of DVT/PE
  * - known May-Thurner Syndrome
* Subject who, in the opinion of the investigator, is not an appropriate candidate for the study

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Blood Velocity | baseline, +10 minutes
  Blood Velocity (Baseline, Peak) will be assessed via ultrasound in the popliteal and femoral veins.
Time Average Mean Velocity | baseline, +10 minutes
  Time Average Mean Velocity (Baseline, Augmented) will be assessed via ultrasound in the popliteal and femoral veins.

SECONDARY OUTCOMES:
Total Volume Flow | baseline, +10 minutes
  Total Volume Flow (Baseline, Augmented) will be assessed via ultrasound in the popliteal and femoral veins.

CONTACTS AND LOCATIONS:
Overall Officials: Fedor Lurie, Principal Investigator — Jobst Vascular Institute
Locations (1):
- Jobst Vascular Institute, Toledo, Ohio, United States

IPD SHARING:
Plan to Share IPD: No